CLINICAL TRIAL: NCT01223586
Title: Extended Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome
Acronym: Ex JAPAN-ACS
Status: Completed | Type: Observational
Sponsor: Kyoto University (Other)
Collaborators: Yamaguchi University Hospital (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University
Organization: Kyoto University Hospital (Other)
Other Study IDs: H22-42
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Statin; Coronary Plaque; Acute Coronary Syndrome; Intravascular Ultrasound; Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regression: Patients with regression of plaque volume by statin
- Non regression: Patients without regression of plaque volume by statin

SUMMARY:
The objective of this study is to verify the relationship between coronary plaque regression and cardiovascular prevention in long term follow up of the Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome (JAPAN-ACS) study [NCT00242944]. In addition, the effect of serum lipid levels or different type of statins on cardiovascular prevention will also be examined.

DETAILED DESCRIPTION:
Several previous multicenter studies using intravascular ultrasound (IVUS) imaging have revealed that statins attenuate the progression of atherosclerosis or even provide regression of plaque volume. Indeed, the Japan Assessment of Pitavastatin and Atorvastatin in Acute Coronary Syndrome (JAPAN-ACS) trial [NCT00242944] has revealed that early aggressive statin therapy in patients with acute coronary syndrome (ACS) significantly reduces the plaque volume of non-culprit coronary lesions On the other hands, a direct relationship between atheroma progression and regression on IVUS and clinical events has not been clearly defined. To verify that relationship, long term follow up of the JAPAN-ACS study will be performed. Clinical outcome of patients with regressed plaque and progressed plaque will be compared. In addition, the objectives of this study are to evaluate the effect of serum lipid levels or different type of statins on cardiovascular prevention.

ELIGIBILITY:
At the enrollment of original study

Inclusion Criteria:

* Patients with written consent by their own volition after being provided sufficient explanation for their participation in this clinical trial
* Patients 20 years or older at the time of their consent
* Patients with hypercholesterolemia as defined by any of the following criteria:

TC >= 220 mg/dL; LDL-C >= 140 mg/dL; Cholesterol-lowering treatment is necessary in accordance with the investigator's judgement when LDL-C >= 100 mg/dL or TC >= 180 mg/dL.

* Patients who have been diagnosed with acute coronary syndrome
* Patients with successful percutaneous coronary intervention (PCI) by intravascular ultrasound (IVUS) guidance
* Patients having coronary plaques (>= 500 µm in thickness or 20% or more in % plaque) at >= 5 mm from the previously treated area in the same branch of coronary artery

Exclusion Criteria:

* Patients with bypass graft or in-stent restenosis at the site of PCI
* Patients who had received PCI on the lesion in the past where the evaluation of coronary plaque volume is planned
* Patients who had plaques in a non-culprit site and might receive PCI during the treatment period
* Patients receiving lipid-lowering drugs (statins, fibrates, probucol, nicotinic acid or cholesterol absorption inhibitors)
* Patients with familial hypercholesterolemia
* Patients with cardiogenic shock
* Patients receiving cyclosporine
* Patients with any allergy to pitavastatin or atorvastatin
* Patients with hepatobiliary disorders
* Pregnant women, women suspected of being pregnant, or lactating women
* Patients with renal disorders or undergoing dialysis
* Patients who are ineligible in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of participants of JAPAN-ACS trial who completed the study
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Composite endpoint | 4-year
  Occurrence of one of following events:
  Cardiovascular death (death from cardiac cause or stroke or peripheral artery disease) Non-fatal Myocardial Infarction (MI) Non-fatal Cerebral Infarction (CI) except for transient ischemic attack (TIA) Unstable angina requiring urgent hospitalizations

SECONDARY OUTCOMES:
Composite cardiovascular events | 4-year
  Occurrence of one of following events:
  Cardiovascular death Non-fatal MI Non-fatal CI Unstable angina requiring hospitalizations Ischemia-driven coronary revascularization except target lesion revascularization (TLR)
Composite coronary heart disease events | 4-year
  Occurrence of one of following events:
  Coronary heart disease (CHD) death Non-fatal MI Unstable angina requiring urgent hospitalizations Ischemia-driven coronary revascularization except TLR
Composite cerebrovascular events | 4-year
  Occurrence of one of following events:
  Fatal and Non-fatal stroke Transient ischemic attack requiring hospitalizations
Mortality | 4-year
  Occurrence of each following events:
  All-cause mortality Cardiovascular death Cardiac death (death from coronary disease or heart failure or arrhythmia and sudden death) CHD death (death from myocardial infarction and sudden death)
Heart disease events | 4-year
  Occurrence of each following events:
  Fatal and Non-fatal MI Non-procedure related MI Procedure related MI Unstable angina requiring urgent hospitalizations Resuscitated cardiac arrest Hospitalization for heart failure PCI or CABG
  1. All events of PCI or CABG
     1. TLR
     2. non-TLR
  2. Ischemia-driven PCI or CABG
     1. TLR
     2. non-TLR
Cerebrovascular events | 4-year
  Occurrence of each following events:
  Fatal and Non-fatal stroke Fatal and Non-fatal CI
  1. Non-procedure related CI
  2. Procedure related CI Fatal and Non-fatal cerebral hemorrhage Hospitalization for TIA
Other events | 4-year
  Occurrence of each following events:
  Operation for or rupture of aortic aneurysm Revascularization for peripheral arterial disease (PAD) Carotid artery stenting (CAS) or carotid endarterectomy (CEA) Aortic dissection Deep vein thrombosis (DVT) or pulmonary thromboembolism (PTE) New occurrence of malignant tumor Operation for aortic stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Masunori Matsuzaki, MD, PhD, Principal Investigator — Professor of Division of Cardiology, Department of Medicine and Clinical Science, Yamaguchi University Graduate School of Medicine
Locations (2):
- Japan (2):
  - Division of Cardiology, Kyoto University Hospital, Kyoto, Kyoto
  - Division of Cardiology, Department of Medicine and Clinical Science, Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi

REFERENCES:
- [Result] Miyauchi K, Daida H, Morimoto T, Hiro T, Kimura T, Nakagawa Y, Yamagishi M, Ozaki Y, Kadota K, Kimura K, Hirayama A, Kimura K, Hasegawa Y, Uchiyama S, Matsuzaki M; JAPAN-ACS Investigators. Reverse vessel remodeling but not coronary plaque regression could predict future cardiovascular events in ACS patients with intensive statin therapy--the extended JAPAN-ACS study. Circ J. 2012;76(4):825-32. doi: 10.1253/circj.cj-12-0135. PMID 22451449